CLINICAL TRIAL: NCT05505539
Title: Intralesional 5-fluorouracil Injection for the Treatment of Oral Leukoplakia: a Pilot Study
Brief Title: Intralesional 5-fluorouracil Injection for the Treatment of Oral Leukoplakia
Acronym: OL_5FU
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator no longer with university.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OL_5FU; 22-36039 (Other: University of California, San Francisco)
Record Dates: First submitted 2022-06-06; First posted 2022-08-17 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5-fluorouracil (Experimental): Participants will receive up to 3 intralesional 5-fluorouracil injections (0.25 mL of a 50mg/mL solution) once every 2 weeks into an oral leukoplakia lesion.
  Interventions: Drug: 5-fluorouracil

INTERVENTIONS:
Drug: 5-fluorouracil — Given intralesionally by injection
  Other Names: 5FU

SUMMARY:
This is a single center, open-label, interventional pilot study to assess the feasibility, safety, and preliminary efficacy of intralesional 5-FU injections for the treatment of oral leukoplakia (OL).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of intralesional 5-fluorouracil (5-FU) injection for the treatment of oral leukoplakia

SECONDARY OBJECTIVE:

I. Evaluate the safety profile and side effects of the study drug.

OUTLINE:

Participants diagnosed with OL will receive multiple intralesional injections of 5-FU solution over a maximum period of 6 weeks, followed by a follow-up visit after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older
* Any gender, race, or ethnicity
* Clinical diagnosis of oral leukoplakia and biopsy proven dysplasia (any grade)
* Oral leukoplakia at least 1 cm in largest diameter
* Ability to understand and willingness to sign a written informed consent document
* Willingness to provide blood and tissue from diagnostic biopsies
* Any smoking history is permitted

Exclusion Criteria:

* Pregnant or lactating women
* Men and women unwilling to use contraception while on study
* History of malignancy that required cytotoxic chemotherapy within the previous 3 months
* Use of 5-FU (systemic or topical) within 3 months prior to study enrollment
* History of allergic reaction or severe hypersensitivity to 5-FU and/or lidocaine
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants s who complete 5-FU injections | Up to 6 weeks
  The number of participants who completed the full course of 3 intralesional injections will be compared to the overall total of participants. If the the mucosa becomes ulcerated or participants are unable/unwilling to continue with therapy, 5FU injections will be stopped.
Number of participants with treatment-related adverse events | Up to 3 months
  The number of participants with documented treatment-related adverse events classified by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported

SECONDARY OUTCOMES:
Change in area of clinically visible oral leukoplakia lesions | Up to 3 months
  The total change in area (measured to nearest millimeter (mm) of clinically visible oral leukoplakia lesion will be defined by the product of the two largest perpendicular measurements. The two largest perpendicular measurements of the treated oral leukoplakia lesion will be measured and multiplied to calculate the lesion area at baseline and again at 3 months.
Proportion of participants with a change in histologic grade | Up to 3 months
  A board-certified oral and maxillofacial pathologist will review biopsy specimens obtained from the treated oral leukoplakia before and after treatment with 5FU and determine change in histologic grade from baseline.
Change in scores on the oral mucosal diseases quality of life questionnaire (COMD-QLQ) | Up to 3 months
  The oral mucosal diseases quality of life questionnaire (COMD-QLQ) is a validated instrument that will assesses the effect that oral leukoplakia has on participants' daily life activities before and after 5-FU intralesional therapy. The survey consists of 24 questions with five response options per item. The response for each item is coded from 0 to 4 with "not at all=0" and "extremely=4" (at time of scoring, for 3 questions, the Likert scale is reversed). The summary of the overall score ranges from 0 to 104, with a higher score indicating a poorer patient-assessed quality of life score.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Jones, DDS, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No